CLINICAL TRIAL: NCT06982547
Title: Clinical Study on the Treatment of Refractory Moderate - to - Severe Active Rheumatoid Arthritis With UTAA91 Injection
Brief Title: Clinical Study on the Treatment of Refractory Rheumatoid Arthritis With UTAA91 Injection
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-011-9
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: UTAA91 injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UTAA91 injection (Experimental)
  Interventions: Biological: UTAA91 injection

INTERVENTIONS:
Biological: UTAA91 injection — After signing the informed consent form, eligible subjects will receive an infusion of UTAA91 injection. Blood samples will be collected from the subjects before and after the infusion for the evaluation of pharmacokinetics, pharmacodynamics, immunogenicity, and safety.

SUMMARY:
This clinical trial is designed as a single - arm, open - label, single - center, investigator - initiated early - phase clinical study. The primary objective is to evaluate the safety of UTAA91 injection in treating subjects with refractory moderate - to - severe active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years (inclusive of the boundary value), with no restriction on gender.
* Expected survival time of at least 3 months.
* Subjects with refractory moderate - to - severe active rheumatoid arthritis who have failed standard treatment or lack effective therapeutic options.
* Meet the requirements for liver and kidney function, as well as cardiopulmonary function.
* Free from severe psychiatric disorders.
* Able to understand the trial and have signed the informed consent form.

Exclusion Criteria:

* A history of malignant tumors other than relapsed/refractory autoimmune diseases (R/R AID) within 5 years prior to screening.
* Subjects with positive results in virus/syphilis tests.
* Severe cardiac diseases or unstable systemic diseases.
* Active or uncontrollable infections requiring systemic treatment within 7 days before administration; evidence of central nervous system invasion at screening.
* Pregnant or breastfeeding women, female subjects planning to become pregnant within 2 years after cell infusion, or male subjects whose partners plan to become pregnant within 2 years after their cell infusion.
* Subjects who have received CAR - T therapy or other gene - modified cell therapies before screening.
* Subjects who participated in other clinical studies within 1 month before screening.
* Other conditions deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2040-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events | About 1 year
  The types, frequency, and severity of adverse events (AEs) and laboratory abnormalities (according to the Common Terminology Criteria for Adverse Events, NCI CTCAE 5.0).

SECONDARY OUTCOMES:
Cmax | About 1 year
  Maximum concentration of UTAA91 injection amplified in peripheral blood after administration of the drug
Tmax | About 1 year
  Time to reach maximum concentration in peripheral blood after administration of UTAA91 injection
Disease remission rate | About 3 months
  The disease remission/response/improvement rates at 28 days, 2 months, and 3 months after treatment with UTAA91 injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No